CLINICAL TRIAL: NCT03175913
Title: Ocoolant Spray vs Lidocaine Infiltration for Reducing the Pain of Spinal Needle Insertion During the Caudal Epidural Injection
Brief Title: Vapocoolant Spray for Reducing the Pain of Spinal Needle Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Collaborators: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Young Eun Moon, associate professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201406018
Record Dates: First submitted 2017-05-30; First posted 2017-06-05 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Vapocoolant spray group (Experimental): vapocoolant spray was applied for 10 second
  Interventions: Device: vapocoolant spray
- Local infiltration group (Active Comparator): 3 ml of 2% lidocaine infiltrated subcutaneously
  Interventions: Drug: local infiltration

INTERVENTIONS:
Device: vapocoolant spray — As a topical pre caudal epidural block anesthesia, spinal needle insertion site was sprayed using an vapocoolant spray for 10-sec from a distance of 30 cm
  Arms: Vapocoolant spray group
Drug: local infiltration — As a topical pre caudal epidural block anesthesia, spinal needle insertion site was injected subcutaneously using 3ml of 2% lidocaine
  Arms: Local infiltration group

SUMMARY:
This was a single-blind, randomized controlled trial. Sixty-six patients who underwent caudal epidural injection were randomized into the vapocoolant spray group or local infiltration group. Before the insertion of a 20-gauge spinal needle, the subcutaneous tissue was infiltrated with 3 ml of 2% lidocaine in the local infiltration group and vapocoolant spray was applied just before the spinal needle insertion in the spray group. 100-mm visual analog scale to evaluate the pain intensity of spinal needle insertion and a five-point Likert scale for patient satisfaction and preference for repeated use were compared between the two groups.

DETAILED DESCRIPTION:
Interventions The intervention room was divided into two sections (intervention section and waiting section) using a blinded partition, for prompt coming and going by the investigators. Before the CEI, patient was informed about how to use a VAS and a five-point Likert scale. Then, patient anxiety about CEI was measured using the Likert scale with the following statement: "I am anxious about undergoing a CEI". After that, the patient was positioned on the table in a prone posture, and the interventionist, who was blinded to the other study procedures, palpated the sacral hiatus and marked with an indelible pen. Then he went behind the partition.

Thereafter, the principal investigator entered the intervention section, opened and checked the sealed envelope. And he prepared the sacrococcygeal area using an iodine-based povidone and an alcohol swabs. As a topical pre-CEI anesthesia, the marked site was infiltrated subcutaneously with 3 ml of 2% lidocaine in the local infiltration group. In the spray group, the marked site was sprayed using an vapocoolant spray (Walter Ritter GmbH and Co., Hamburg, Germany) for 10-sec from a distance of 30 cm. To enhance a blind design, 10-sec spray was performed with targeting to the open air after 3 min (time for manifesting the effect of lidocaine) in the local infiltration group. In the spray group, there had been same time interval of 3 min before spraying.

Immediately after these procedures, the marked site was prepped again using alcohol swab, then the principal investigator left and the interventionist entered the intervention section. And the interventionist inserted a prepared 20-gauge spinal needle into the marked site and pointed the needle toward the sacral hiatus under ultrasonography (Xario, Toshiba, Otawara, Japan) guided. When neither tissue resistance nor subcutaneous injection was noticed after injecting saline, 15 ml of 0.5% lidocaine and 10 mg of dexamethasone were injected.

After finishing the CEI, each patient was asked to fill out the self-administered documents for outcome measures, seal them in an envelope, and submit them to the principal investigator.

Outcome Measures Pain induced by spinal needle insertion was assessed using a 100-mm VAS as well as patients' satisfaction about the topical pre-CEI anesthesia using a five-point Likert scale. The 100-mm VAS consisted of a 100-mm horizontal line labeled "no pain" at the left and "worst pain imaginable" at the right. The five-point Likert scale (1, strongly agree; 2, agree; 3, undecided; 4, disagree; and 5, strongly disagree) was used to answer two questions: ''Are you satisfied with the topical pre-CEI anesthesia used before the spinal needle insertion of CEI?'' and ''Will you use the topical pre-CEI anesthesia applied today again if CEI repeated in the future?''

ELIGIBILITY:
Inclusion Criteria:

* patients with low back pain and radiating pain in the lower limb who underwent a scheduled caudal epidural injection

Exclusion Criteria:

* those who had systemic inflammatory disease, those who take anticoagulant administration, those who had uncontrolled diabetes, those who were unable to understand a visual analog scale (VAS) or a Likert scale, those with a history of cold intolerance or cold allergy, those with a history of allergic reaction to lidocaine, those who took pain medications or had used topical anesthetics within the previous 24 hrs, those who had a skin lesion on the sacral hiatus, and those who had the experience of caudal epidural injection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
100mm visual analog scale | Up to 20 minutes (Just after caudal epidural injection)
  Pain of spinal needle insertion during caudal epidural injection

SECONDARY OUTCOMES:
Five point Likert scale | Up to 20 minutes (Just after caudal epidural injection)
  five-point Likert scale (1, strongly agree; 2, agree; 3, undecided; 4, disagree; and 5, strongly disagree) was used to answer two questions: ''Are you satisfied with the topical pre-CEI anesthesia used before the spinal needle insertion of CEI?'' and ''Will you use the topical pre-CEI anesthesia applied today again if CEI repeated in the future?''

IPD SHARING:
Plan to Share IPD: No